CLINICAL TRIAL: NCT07220681
Title: A Hybrid I Evaluation of Integrative Health Care for PTSD
Brief Title: Integrated Health Care for PTSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HT94252510881
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: PTSD; complementary and integrative health; Veterans; implementation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Yoga; Meditation; Health

STUDY DESIGN:
Intervention Model Description: * Hybrid Type 1 study, simultaneously assessing efficacy and gathering information relevant to implementation
  * "Drop the loser" adaptive design, whereby any experimental condition lagging behind the other conditions will be discontinued after interim analysis
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual care (Active Comparator): Information about local and national complementary and integrative health programs
  Interventions: Other: Information
- Yoga and meditation (Experimental): Hatha yoga classes via videoconferencing and self-learning of Mantram Repetition Program
  Interventions: Behavioral: Yoga and meditation; Other: Information
- Wellness (Experimental): Weekly exercise/nutrition classes to support lifestyle changes
  Interventions: Behavioral: Wellness; Other: Information
- Positive affect (Experimental): Weekly classes focused on increasing positive affect and social support
  Interventions: Behavioral: Positive affect; Other: Information

INTERVENTIONS:
Behavioral: Yoga and meditation — 12 weekly 60-minute hatha yoga classes and access to video-based training in a portable mantra-based meditation practice
  Arms: Yoga and meditation
Behavioral: Wellness — 12 weekly 60-minute classes to provide education about exercise and nutrition and facilitate lifestyle changes
  Arms: Wellness
Behavioral: Positive affect — 12 weekly 60-minute classes to teach strategies for increasing positive affect and to provide social connection
  Arms: Positive affect
Other: Information — Provision of written information about local and national complementary and integrative care resources

SUMMARY:
The goal of this clinical trial is to determine whether which types of integrative care, meaning a combination of psychotherapy and mind-body interventions, lead to the most changes in functioning among Veterans with posttraumatic stress disorder (PTSD). The main aims are:

1. To evaluate the impact of integrative care approaches on functional outcomes among Veterans with PTSD.
2. To examine factors relevant to the implementation of integrated treatments for PTSD from the perspective of patients, providers and administrators in the VA Healthcare System.

Participants will:

1. Complete assessments at the beginning of the study and 12- and 24-weeks later.
2. Engage in 12 weeks of integrated care, with the type being randomly assigned.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis
* eligibility for Cognitive Processing Therapy (CPT) at a participating VA site
* able to consent to study activities

Exclusion Criteria:

* current, active engagement in one of the included approaches (per clinician judgment)
* medical conditions that contraindicate engaging in the experimental interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Inventory of Psychosocial Functioning (IPF) | weeks 0, 12 and 24
  The IPF is a self-report measure of functioning across several domains. It is summarized in a mean score with higher scores indicating greater functional impairment.

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 Revised (CAPS-5R) | weeks 0, 12 and 24
  The CAPS-5R is a clinician-administered measure of PTSD symptom severity summarized in a total score with higher scores indicating greater symptom severity.
Quick Inventory of Depressive Symptomatology (QIDS) | weeks 0, 12 and 24
  The QIDS is a self-report measure of depression severity summarized by a total score for which higher scores reflect greater symptom severity.
Insomnia Severity Index (ISI) | weeks 0, 12 and 24
  The ISI is a self-report measure that assesses the consequences of and distress related to insomnia summarized by a total score in which higher scores indicate greater sleep disruption.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - VA Central Arkansas Healthcare System, Little Rock, Arkansas
  - VA San Diego Healthcare System, San Diego, California
  - VA Portland Healthcare System, Portland, Oregon
  - VA North Texas Healthcare System, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Deidentified datasets will be made available via National Institutes of Mental Health Data Archive (NDA). The study protocol, statistical analysis plan and ICF/HIPAA form will be available on clinical.trials.gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data and supporting information will be available within 1 year of the conclusion of the trial and archived according to the standards of the hosting archives.
Access Criteria: Unique research resources will be readily available for research purposes to members of academic institutions, non-profit organizations, and commercial partners after the completion of data analysis, presentations, and publications
URL: https://nda.nih.gov/